CLINICAL TRIAL: NCT03173820
Title: Clinical Trial in Assigning of Tacrolimus Dosage Regimen According to CYP3A5 Genotype in Kidney Transplant Recipients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Collaborators: National Science and Technology Development Agency, Thailand (Other Government)
Responsible Party: Principal Investigator, Suda Vannaprasaht, Department of Medicine, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KhonKaenU_tacrolimus
Record Dates: First submitted 2017-05-22; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-06

CONDITIONS: Kidney Transplantation
Keywords: tacrolimus; transplantation; CYP3A5; genotype
MeSH Terms: interventions — Congresses as Topic

STUDY DESIGN:
Intervention Model Description: genotype guided vs conventional tacrolimus dosage regimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Conventional (Placebo Comparator): no genotype of CYP3A5 investigated to adjust tacrolimus dosage regimen
  Interventions: Genetic: Conventional
- Genotype guided (Active Comparator): Use CYP3A5 genotype to adjust dosage regimen for tacrolimus
  Interventions: Genetic: Genotype guided

INTERVENTIONS:
Genetic: Genotype guided — Tacrolimus will be prescribed depend on CYP3A5 genotype. CYP3A5*1/*1 patients will receive tacrolimus 0.125 mg/kg/day. CYP3A5*1/*3 patients will receive tacrolimus 0.1 mg/kg/day. CYP3A5*3/*3 patients will received tacrolimus 0.08 mg/kg/day. Tacrolimus target level for this phase will be 5-8 ng/ml.
  Arms: Genotype guided
Genetic: Conventional — Tacrolimus will be prescribed 0.1 mg/kg /day for all patients to achieve tacrolimus level 5-8 ng/ml.
  Arms: Conventional

SUMMARY:
Kidney transplantation is the most appropriated treatment in end stage renal failure patients in order to improve quality of life. However, patients have to take immunosuppressive drugs to prevent graft rejection. Tacrolimus is the most common immunosuppressive drug used now. However, tacrolimus has narrow therapeutic level and needs regularly therapeutic monitor because of inter-individual variation in dosage regimen. Not only age, body weight and drug interaction but also genetic factor in metabolic pathway of tacrolimus plays an important role in tacrolimus blood level. Previous data showed CYP3A5 genetic polymorphism was significant effect tacrolimus blood level. From previous study showed the mean dose of tacrolimus required for the induction phase was significantly higher (P= 0.006) in the CYP3A5*1/*1 group at 0.142±0.050 mg/kg/day than that required by patients who carried either the CYP3A5*1/*3 group of 0.097±0.040 mg/kg/day or the CYP3A5*3/*3 group of 0.077±0.020 mg/kg/day. Tacrolimus maintenance dose required for CYP3A5*1/*1 group of 0.12±0.03 mg/kg/day was 1.3 times higher (P<0.0001) than used for the CYP3A5*1/*3 at 0.09±0.03 mg/kg/day and 2.4 times higher than the CYP3A5*3/*3 group of 0.05±0.02 mg/kg/day. Therefore, the investigators plan to investigate a prospective study to determine the clinical outcome of tacrolimus treatment in kidney transplant recipients between genotype guided dosage regimen group and conventional group.

DETAILED DESCRIPTION:
Objective

1. To determine the clinical outcome of tacrolimus treatment in kidney transplant recipients between genotype guided dosage regimen group and conventional group
2. To determine the influence of CYP3A5 polymorphism on clinical outcome of kidney transplantation recipients Review article Kidney transplantation is the most appropriated treatment in end stage renal failure patients in order to improve quality of life. National health security office of Thailand estimates the cost of kidney transplantation around 250,000 to 400,000 baht per patient. However, patients have to take immunosuppressive drugs such as cyclosporine, tacrolimus, azathioprine, mycophenolate, prednisolone etc. to prevent graft rejection. Tacrolimus is a common immunosuppressive drug used worldwide. However, tacrolimus has narrow therapeutic level and needs regularly therapeutic monitor because of inter-individual variation in dosage regimen. Achieving and maintaining target concentration of tacrolimus are related to tacrolimus toxicity and graft rejection. Not only age, body weight and drug interaction but also genetic factor in metabolic pathway of tacrolimus plays an important role in tacrolimus blood level.

Cytochrome P450 3A4 (CYP3A4) and CYP3A5 are the main enzyme responsible for metabolism of tacrolimus. Unlike CYP3A4, CYP3A5 is more polymorphic and expression of enzyme is controlled by CYP3A5 gene variants. CYP3A5*3, an A to G transition (A6986G) within intron 3 results in the production of a truncated protein, is the most common allele variant. From previous study of our group, the allele frequency of CYP3A5*3 was 66% which is lower than those reported in the Caucasian population (85%). Prevalence of CYP3A5*1/*1, CYP3A5*1/*3, CYP3A5*3/*3 in 400 healthy Thai volunteers are 13.75%, 42.75% and 43.50%, respectively (unpublished data).

Patients who carried CYP3A5*1/*1 or CYP3A5*1/*3 allele showed tacrolimus clearance higher than CYP3A5*3/*3 patients (0.679 ± 0.195 vs 0.355 ± 0.091 L/h/kg). Therefore, CYP3A5*3/*3 patients received 48% lower dose of tacrolimus than CYP3A5*1/*1 or CYP3A5*1/*3 patients in order to achieve the same therapeutic range.

From our previous study showed the mean dose of tacrolimus required for the induction phase was significantly higher (P= 0.006) in the CYP3A5*1/*1 group at 0.142±0.050 mg/kg/day than that required by patients who carried either the CYP3A5*1/*3 group of 0.097±0.040 mg/kg/day or the CYP3A5*3/*3 group of 0.077±0.020 mg/kg/day. Tacrolimus maintenance dose required for CYP3A5*1/*1 group of 0.12±0.03 mg/kg/day was 1.3 times higher (P<0.0001) than used for the CYP3A5*1/*3 at 0.09±0.03 mg/kg/day and 2.4 times higher than the CYP3A5*3/*3 group of 0.05±0.02 mg/kg/day.

Previous prospective randomized study showed higher proportion of patients who received genotype guided tacrolimus dosage regimen had achieved the target blood level at day 3 after started tacrolimus than control group. This study did not show difference clinical outcome between two groups and follow period was short, only three months. This study investigated only in induction phase.

Because most of studies investigated only in induction phase and follow up period was short. The present study will conduct a randomized prospective study to evaluate whether adaption of tacrolimus dosing according to CYP3A5 genotype in both induction and maintenance phase after transplantation can achieve target concentration than control group. Moreover, the present study will investigate the influence of CYP3A5 polymorphism on kidney transplant outcome.

Methods This prospective, open label, randomized study will conduct at Nephrology Unit, Department of Medicine, Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand. This study was approved by Khon Kaen University Research Ethics Committee for Human Research, Khon Kaen University, Thailand (HE551389)

The patients will randomly assigned to receive tacrolimus at either a fixed dosage (conventional group) or genotype guided dosage group.

1. Induction Phase (0-4 weeks) Patients who will be assigned in conventional group will receive tacrolimus 0.1 mg/kg /day. Patients who will be in genotype guided group, will receive tacrolimus depend on CYP3A5 genotype. CYP3A5*1/*1 patients will receive tacrolimus 0.125 mg/kg/day. CYP3A5*1/*3 patients will receive tacrolimus 0.1 mg/kg/day. CYP3A5*3/*3 patients will receive tacrolimus 0.08 mg/kg/day. Tacrolimus target level for this phase will be 5-8 ng/ml.
2. Maintenance Phase (5-24 weeks) Patients who will be in conventional group, will receive tacrolimus 0.08 mg/kg/day. Patients who will be in genotype guided group, will receive tacrolimus depend on CYP3A5 genotype. CYP3A5*1/*1 patients will receive tacrolimus 0.12 mg/kg/day. CYP3A5*1/*3 patients will receive tacrolimus 0.08 mg/kg/day. CYP3A5*3/*3 patients will receive tacrolimus 0.04 mg/kg/day. Tacrolimus target level for this phase will be 3-5 ng/ml.

Patients will randomized prior to transplantation according to block of four computer generate randomization. The patients will followed for 6 months unless they will be withdrawn from the study or lost follow up Inclusion criteria Kidney transplantation recipients who

1. Age > 18 year old
2. Will have kidney transplantation at Srinagarind hospital, Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand
3. Will have the first kidney transplantation
4. Will receive tacrolimus as immunosuppressive to prevent graft rejection
5. Will have aspartate transaminase and alanine transaminase < 2 time of normal level, total bilirubin <1.5 mg/dl and direct bilirubin within normal limited
6. Welling to be volunteer in this study and sign the inform consent Exclusion criteria Kidney transplantation recipients who

1. Refuse to join this study 2. Have history of drug allergy to tacrolimus 3. Is pregnancy and lactating Intervention All renal transplantation waiting list patients will invited to join this study and sign inform consent. The patients who will be enroll to this study, will be drawn the blood for 6 ml to perform CYP3A5 genotype assay.

Patients who perform kidney transplantation and enrolled to this study will randomly assign in equal number to receive tacrolimus doses as in table 1, one hour before transplantation and after transplantation. Tacrolimus blood level, blood urea nitrogen (BUN)/creatinine (Cr), will regularly perform on day 1, 3, 4, 5, 7, 14 and 28 during induction phase (1st-4th week after kidney transplantation). Moreover, urine 24 hour for Cr, protein will perform in day 7, 14, 28 after transplantation. The physicians will modify the daily dose of tacrolimus according to their practice in order to achieve target range of trough concentration (5-8 ng/ml). Patients will receive other immunosuppressive such as corticosteroid, mycophenolate mofetil as general practice.

During maintenance phase (5th-24th week after kidney transplantation) tacrolimus doses will be adjusted as in table 1. Tacrolimus blood level, BUN/Cr and urine 24 hour for Cr and protein will be perform on 5, 8, 12, 16, 20, 24 after transplantation. The physicians will modify the daily dose of tacrolimus according to their practice in order to achieve target range of trough concentration (3-5 ng/ml).

DNA extraction and genotype Peripheral blood samples will collect from individual subjects. Genomic DNA sample will be extracted from buffy coat by QIAamp® DNA Blood Mini kit. CYP3A5 genotype will be examined by Real-time polymerase chain reaction (Real-time PCR). Analysis of CYP3A5*3 will be performed using Custom TaqMan® Single nucleotide polymorphism Genotyping Assay (Applied Biosystem, Foster city, California) on an ABI PRISM® 7500 Real-Time PCR System (Applied Biosystem, Foster city, California). In brief, 25 μl of reaction mixtures will consist of 100 ng of genomic DNA, TaqMan® Universal PCR Master Mix and TaqMan® MGB primers and specific CYP3A5*3 probes. The sense primer will be 5'- CGAATGCTCTACTGTCATTTCTAACCA -3' and the antisense primer will be 5'- TGAAGGGTAATGTGGTCCAAACAG -3'. The CYP3A5*1 probe was 5'- TTTGTCTTTCAATATCTC -3' labeled with 6-carboxyfluorescein (FAM) and the CYP3A5*3 probe will be 5'- TTTGTCTTTCAGTATCTC -3' labeled with 50-fluorescein (VIC). The reaction mixtures will be incubated at 50oC for 2 min for AmpErase® Uracil N-Glycosylase (UNG). UNG degradation of any carryover DNA contamination, followed by AmpliTaq® Gold enzyme activation at 95 degree Celsius for 10 min. Amplification will be performed for 40 cycles in which each cycle consisted of denaturation at 92 degree Celsius for 15 sec will follow by annealing and primer extension at 60 degree Celsius for 1 minute. The real time PCR base sequences will be confirmed by gene sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplantation recipients who

  1. Age > 18 year old
  2. Will have kidney transplantation at Srinagarind hospital, Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand
  3. Will have the first kidney transplantation
  4. Will receive tacrolimus as immunosuppressive to prevent graft rejection
  5. Will have AST and ALT < 2 time of normal level, total bilirubin <1.5 mg/dl and direct bilirubin within normal limited
  6. Welling to volunteer in this study and sign the inform consent

Exclusion Criteria:

* Kidney transplantation recipients who

  1. Refuse to join this study
  2. Have drug allergy to tacrolimus
  3. Have Pregnancy and lactating Intervention All renal transplantation waiting list patients will invited to join this study and sign inform consent. The patients who will be enroll to this study, will be drawn the blood for 6 ml to perform CYP3A5 genotype assay.

Patients who perform kidney transplantation and enrolled to this study will randomly assign in equal number to receive tacrolimus doses as in table 1 hr before transplantation and after transplantation. Tacrolimus blood level, BUN/Cr, will regularly perform on day 1, 3. 4, 5, 7, 14 and 28 during induction phase (1st-4th week after kidney transplantation). Moreover, urine 24 hour for Cr, protein will perform in day 7, 14, 28 after transplantation. The physicians will modify the daily dose of tacrolimus according to their practice in order to achieve target range of trough concentration (5-8 ng/ml). Patients will receive other immunosuppressive such as corticosteroid, mycophenolate mofetil as general practice.

During maintenance phase (5th-24th week after kidney transplantation) tacrolimus doses will be adjusted as in table 1. Tacrolimus blood level, BUN/Cr and urine 24 hour for Cr and protein will be perform on 5, 8, 12, 16, 20, 24 after transplantation. The physicians will modify the daily dose of tacrolimus according to their practice in order to achieve target range of trough concentration (3-5 ng/ml).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-04-30 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean tacrolimus level | at day 3 after transplantation
  Proportion of patients whose tacrolimus level were in therapeutic range at day 3 post transplantation

SECONDARY OUTCOMES:
Mean tacrolimus level | at day 1, 3, 5, 7, 14, 30,60, 90, 120, 150 and 180 days post transplantation
  Proportion of patients whose tacrolimus level were in therapeutic range at day 1, 3, 5, 7, 14, 30,60, 90, 120, 150 and 180 days post transplantation
Incidence of delay graft rejection | day 1- 6 month after transplantation
  Compare incidence of delay graft rejection between 2 groups
Mean GFR level | at day 7, 14, 30, 60, 90, 120, 150, and 180 days after transplantation
  Compare mean GFR level at day 7, 14, 30, 60, 90, 120, 150, and 180 days after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Suda Vannaprasaht, MD, Principal Investigator — Faculty of Medicine, Khon Kaen University
Locations (1):
- Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No